CLINICAL TRIAL: NCT07195617
Title: Clinical Study on Evaluating the Safety and Effectiveness of BCMA-GPRC5D CAR-T in Patients With Relapsed/Refractory Multiple Myeloma Who Have Received Third-line or Above Treatment
Acronym: r/r MM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Collaborators: Jiangsu Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG-CT-24-015
Record Dates: First submitted 2025-04-09; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-08

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Subjects signed informed consent voluntarily, and for those who met the inclusion criteria and did not meet the exclusion criteria, intravenous infusion of 2×106 /kg±50% CAR T cells was performed at D0.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCMA-GPRC5D CAR T cells were transfused (Experimental): Subjects voluntarily signed informed consent and were evaluated during blood collection, pre-treatment and pre-transfusion. Eligible subjects received intravenous infusion of 2×106 /kg±50% CAR T cells.
  Interventions: Drug: BCMA-GPRC5D CART

INTERVENTIONS:
Drug: BCMA-GPRC5D CART — The entire study process was as follows: Screening period (V1) : Informed consent was signed, screening was checked, criteria were evaluated, and baseline demographic information and subject status were recorded. Blood collection period (V2) : For subjects who meet the inclusion and exclusion criteria, the blood required for CAR-T preparation will be obtained by leukocyte isolation monopexy or intravenous collection according to the conditions of the subjects. Preconditioning phase (V3) : cytokine and cell changes. Pre-transfusion assessment (V4) : The investigator assessed that the test results met the cell transfusion criteria, and D0 CAR T cell infusion could be performed with investigator permission. Infusion phase (V5) : CAR-T cells were transfused according to the dosage and method specified in the protocol. Safety and efficacy were followed up on D1, D4, D7, D10, D14, D21, D28, M3, M6, M9, M12, and M24.

SUMMARY:
This study is a single-arm, single-center clinical study, with the main purpose of IIT clinical trials to evaluate the safety and initial efficacy of BCMA-GPRC5DCAR-T cells in subjects with relapsed/refractory multiple myeloma (r/rMM). The dose of this study was set to 2.0×106/kg±50% CAR-T cells, and the infusion method was a single peripheral infusion.

After the screening period (W-8~D-8), blood collection period (W-8~D-8), pretreatment period (D-7~D-3), and pre-infusion evaluation (D-2~D-1), subjects were subjected to infusion of CAR-T cells in D0. After administration, they were subjected to safety, effectiveness and other related examinations according to the follow-up plan. The subjects followed up until 2 years after cell re-infusion or the subject met the withdrawal treatment standards, whichever occurs first.

DETAILED DESCRIPTION:
The entire study process was as follows: Screening period (V1) : Informed consent was signed, screening was checked, criteria were evaluated, and baseline demographic information and subject status were recorded. Blood collection period (V2) : For subjects who meet the inclusion and exclusion criteria, the blood required for CAR-T preparation will be obtained by leukocyte isolation monopexy or intravenous collection according to the conditions of the subjects. Preconditioning phase (V3) : cytokine and cell changes. Pre-transfusion assessment (V4) : The investigator assessed that the test results met the cell transfusion criteria, and D0 CAR T cell infusion could be performed with investigator permission. Infusion phase (V5) : CAR-T cells were transfused according to the dosage and method specified in the protocol. Safety and efficacy were followed up on D1, D4, D7, D10, D14, D21, D28, M3, M6, M9, M12, and M24. Subjects were followed up to M24 or those who met the exit criteria withdrew early, whichever happened first.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or his/her guardian understands and voluntarily signs informed consent form, and is expected to complete the follow-up examination and treatment of the research procedure;
2. Ages 18-75 years old (including the threshold), gender is not limited;
3. Patients diagnosed with multiple myeloma according to the IMWG diagnostic criteria;
4. Determine that there are measurable lesions during screening according to any of the following criteria: serum single cloned paraprotein (M-protein) level ≥1.0g/dL or urine M-protein level ≥200mg/24 hours; or light chain multiple myeloma diagnosed with serum or urine: serum immunoglobulin free light chain ≥10mg/dL and serum immunoglobulin κ/γ free light chain ratio ;
5. Previously received treatment with at least three-line multiple myeloma;
6. Materials have proved that the patient's multiple myeloma disease is relapse-refractory or primary-refractory, defined as:

   1. relapse-refractory: non-responsive to rescue treatment (no response is defined as the inability to obtain a slight remission [MR] or disease progression in treatment), or disease progression within 60 days of the last treatment, or MR or above remission has occurred;
   2. primary-refractory: patients who have never obtained MR or above treatment, including patients who have never obtained MR or above remission, but have little change in M protein, have no evidence of clinical progress, and are subject to the definition of progress.
7. The patient has recovered from the toxicity of the previous treatment, that is, the CTCAE toxicity grade is < 2 (unless the abnormality is related to the tumor or is judged by the researcher to be in a stable state, and has little impact on safety or efficacy);
8. ECOG physical fitness status score 0 to 1 point and the estimated survival period is greater than 3 months;
9. Have appropriate organ functions:

   1. Alanine aminotransferase (ALT) ≤3 times the upper limit of normal value (ULN);
   2. Alanine aminotransferase (AST) ≤3 times the ULN;
   3. Total bilirubin ≤1.5 times the ULN;
   4. Serum creatinine ≤1.5 times the ULN, or creatinine clearance ≥60mL/min;
   5. Hemoglobin ≥50g/L (no blood transfusion support must be received within 7 days before laboratory examination );
   6. Indoor oxygen saturation ≥92%;
   7. Correction of serum calcium ≤12.5 mg/dL (≤3.1 mmol/L) or free ionic calcium ≤6.5 mg/dL (≤1.6 mmol/L);
   8. Left ventricular ejaculation fraction (LVEF) ≥45%, echocardiography confirms that no pericardial effusion is seen, and no clinically significant electrocardiogram discovery is found;
   9. There is no clinically significant pleural effusion;
10. The venous pathway required for collection can be established, and there are no contraindications for white blood cell collection.

Exclusion Criteria:

1. Diagnosed or treated with other aggressive malignant tumors other than multiple myeloma within 3 years;
2. Previously received anti-tumor treatment (before blood collected for CAR-T preparation): received targeted therapy, epigenetic therapy or experimental drug treatment within 14 days or at least 5 half-life (whichever is shorter) or used for invasive experimental medical devices; treated with monoclonal antibodies within 21 days; received cytotoxic treatment within 14 days; received proteasome inhibitors within 14 days; received immunomodulatory agents within 7 days; received radiotherapy within 14 days (except for 5% bone marrow reserves);
3. Suspected that MM has been involved in the central nervous system or meninges and has been confirmed by magnetic or CT, or has other active central nervous system diseases;
4. Suffered from Fahrenheit macroglobulinemia, POEMS syndrome (multiple neuropathy, enlarged organs, endocrine lesions, monoclonal protein diseases and skin changes) or primary AL amyloidosis during screening;
5. Hepatitis B surface antigen (HBsAg) positive, or hepatitis B core antibody (HBcAb) positive and peripheral blood HBV DNA quantitative test; hepatitis C virus (HCV) antibody positive; human immunodeficiency virus (HIV) antibody positive; cytomegalovirus (CMV) DNA test; EB virus DNA test; syphilis test positive;
6. People with a history of severe allergic allergies [the history of severe allergies is defined as a secondary or above all allergic reaction, and any of the following clinical manifestations appear when an allergic reaction occurs: airway obstruction (running nose, cough, Stirrhage, dyspnea), tachycardia, hypotension, arrhythmia, gastrointestinal symptoms (nausea, vomiting), incontinence, laryngeal edema, bronchospasm, cyanosis, shock, respiratory, cardiac arrest] or known to be allergic to any drug active ingredients, excipients or mouse-derived products or xenoproteins contained in this trial (including the clearing regimen);
7. Suffering from severe heart disease, including but not limited to severe arrhythmia, unstable angina, large-area myocardial insufficiency, New York Heart Association Grade III or IV cardiac insufficiency, myocardial infarction ≤6 months before screening or receiving Coronary artery bypass bypass (CABG), a history of syncope with unknown causes and non-vasovagal or dehydration, a history of severe non-ischemic cardiomyopathy, and refractory hypertension (refractory hypertension is defined as: a sufficient amount of ≥3 antihypertensive drugs (including diuretics) that are reasonably tolerated on the basis of improving lifestyle > 1 month of blood pressure still not meet the standards or taking ≥4 antihypertensive drugs to effectively control blood pressure);
8. Systemic diseases that are unstable by the researchers: including but not limited to severe liver, kidney or metabolic diseases that require drug treatment;
9. Before screening Patients with acute/chronic graft-versus-host disease (GVHD) within 6 months or need to receive immunosuppressants for GVHD;
10. Patients with active nervous system autoimmunity or inflammatory diseases (such as: Guillin-Barre syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular diseases (such as cerebral edema, posterior reversible encephalopathy syndrome (PRES));
11. Patients with emergency tumor emergencies (such as spinal cord compression, intestinal obstruction, leukocyte stasis, tumor lysis syndrome, etc.) that require emergency treatment;
12. There are uncontrollable bacteria, fungi, viruses or other infections that require antibiotic treatment;
13. The screening time has used short-acting hematopoietic cytokine drugs that have an effect on the patient's blood sign within 1 week after the planned blood collection for CAR-T preparation, or long-acting hematopoietic cytokine drugs within 2 weeks, and the researchers have determined that it has an effect on cell preparation.
14. During the screening period, hormone or immunosuppressant drugs are being received within 2 weeks of blood collection planned to prepare CAR-T, and the researchers judged that it has an impact on cell preparation:

    1. Hormones: Subjects who were receiving systemic steroids within 2 weeks of the planned blood collection for CAR-T preparation and who were deemed to require long-term use of systemic steroids during treatment (except inhaled or topical use); and subjects who were using systemic steroids within 72 hours before cell reentering (except inhaled or topical use);
    2. Immunization Inhibitors: Those who are undergoing immunosuppressors within 2 weeks of the planned blood collection for the preparation of CAR-T during screening;
15. Those who have undergone major surgical operations (except diagnostic surgery and biopsy) or major surgery during the study period within 4 weeks before the study period, or those who have not fully healed before the enrollment;
16. Those who have received (attenuated) live virus vaccine within 4 weeks before the screening;
17. Those who have severe mental illness;
18. Those who have alcoholics or have a history of drug abuse;
19. Women who are pregnant or breastfeeding, and female subjects who are planning to pregnancy within 2 years after cell rebirth or male subjects who are planning to pregnancy within 2 years after cell rebirth;
20. Subjects who have contraindications to any research procedure or who have other medical conditions that may put them at unacceptable risks according to the investigator's judgment and/or clinical standards.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint indicator: safety assessment | All AE and SAE were collected after cell reinfusion and recorded until 2 years after subjects withdrew from the study or cell reinfusion, whichever occurs first.
  Safety assessment is carried out for all adverse events and other safety indicators such as laboratory examinations.

SECONDARY OUTCOMES:
Concentration of CAR-T cells after Infusion (PK) | From enrollment to the end of treatment at 24 months
  CAR-T in peripheral blood after infusion
Concentration of Cytokine after Infusion (PD) | Up to 24 months.
  Calculate the change of cytokine concentration in peripheral blood after After CAR-T infusion. Cytokines include IL-2、IL-6 and so on.
overall response rate, ORR | Up to 24 months.

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial, only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code